CLINICAL TRIAL: NCT06106841
Title: A Phase Ib/II Clinical Trial of TQB3909 Tablets in Subjects With Relapsed or Refractory MCL Safety and Efficacy
Brief Title: TQB3909 Tablets in Subjects With Relapsed or Refractory Mantle Cell Lymphoma (MCL)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated for strategic business reasons
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3909-Ib/II-04
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 400mg of TQB3909 tablets (Experimental): tablet, 28 days as a treatment cycle.
  Interventions: Drug: 400mg of TQB3909 tablets
- 600mg of TQB3909 tablets (Experimental): tablet, 28 days as a treatment cycle.
  Interventions: Drug: 600mg of TQB3909 tablets

INTERVENTIONS:
Drug: 400mg of TQB3909 tablets — TQB3909 tablets 400mg, TQB3909 tablets is a B-cell lymphoma (BCL)-2 inhibitor.
  Arms: 400mg of TQB3909 tablets
Drug: 600mg of TQB3909 tablets — TQB3909 tablets 600mg, TQB3909 tablets is a B-cell lymphoma (BCL)-2 inhibitor.
  Arms: 600mg of TQB3909 tablets

SUMMARY:
This is a study to assess the safety of TQB3909 monotherapy in participants with relapsed or refractory MCL.

ELIGIBILITY:
Inclusion Criteria:

* The subject voluntarily joins the study, signs the informed consent form, and has good compliance;
* Age: ≥ 18 years old (when signing the informed consent form); Eastern Cooperative Oncology Group performance status (ECOG PS) score: 0-2 points; Expected survival is more than 3 months;
* Subject population: Confirmed as MCL by local laboratory pathology and independent pathology review (stage 2).
* The main organs are functioning well,
* The patient's Computed Tomography (CT) / Magnetic Resonance Imaging (MRI) shows measurable lesions, defined as ≥ 1 lymph node with the longest diameter of > 1.5 cm or ≥ 1 extranodal lesion with the longest diameter of > 1.0 cm, which can be measured by ≥ 2 vertical dimensions;
* Female subjects of childbearing age should agree to use contraception (e.g., pills, or condoms) during the study and for 6 months after the end of the study; Have a negative serum pregnancy test within 7 days prior to study enrollment and must be a non-lactating subject; Male participants should agree that contraception must be used during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

* Have had or currently have other malignant tumors within 3 years before the first dose of study drug.
* It is known that lymphoma affects the central nervous system (CNS);
* Previous allogeneic hematopoietic stem cell transplantation;
* Have received autologous hematopoietic stem cell transplantation within 3 months before the first dose of study drug;
* There are a variety of factors that affect oral drugs (such as inability to swallow, chronic diarrhea and intestinal obstruction, inflammatory bowel disease, malabsorption syndrome, etc.);
* Unmitigated toxicity ≥ Common Terminology Criteria for Adverse Events (CTCAE) grade 2 due to any prior treatment (except hair loss, absolute neutrophil count and platelet abnormalities, which follow the inclusion criteria 4);
* Significant surgical treatment and obvious traumatic injury within 28 days prior to the start of study treatment;
* Arteriovenous thrombotic events within 3 months before the first dose, such as cerebrovascular accident (including cerebral hemorrhage, cerebral infarction, except lacunar cerebral infarction), deep vein thrombosis (except secondary to deep vein catheterization) and pulmonary embolism;
* Those who have a history of psychotropic substance abuse and cannot be withdrawn or have mental disorders;
* Subjects with any severe and/or uncontrolled medical conditions, including:
* Grade ≥2 myocardial ischemia or myocardial infarction, arrhythmia (Quick Time Constant Fluctuation (QTcF) >450 ms in men, QTcF >470 ms in women) and grade ≥2 congestive heart failure (New York Heart Association (NYHA) grade), cardiac ultrasound assessment of left ventricular ejection fraction (LVEF) of <50%; poorly controlled hypertension, defined as systolic blood pressure > 170 mmHg and diastolic blood pressure > 105 mmHg at least 2 consecutive blood pressure measurements at the time of screening；
* presence of active infection (≥ CTCAE grade 2 infection);
* active hepatitis; Hepatitis B virus (HBV) infection, HBV DNA positive or copy number exceeding the upper limit of normal values in the research center;
* Have a history of immunodeficiency, including Human Immunodeficiency Virus(HIV)-positive or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
* Those who have epilepsy and need treatment.
* Have received chemotherapy and radiotherapy within 4 weeks before the first dose, received immune checkpoint inhibitors and Chimeric Antigen Receptor T-Cell Immunotherapy (CAR-T) therapy 12 weeks before the first dose, and received other small molecule antitumor therapy (elution period from the end of the last treatment) before the first drug use within 5 half-lives;
* Previous treatment with BCL-2 inhibitors;
* Have received a live vaccine within 4 weeks prior to the first dose, or plan to be vaccinated during the study;
* Have participated in other antitumor drug clinical trials within 4 weeks before the first dose;
* According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of subjects or affect the completion of the study, or subjects who are considered to be unsuitable for enrollment for other reasons.
* Allergic to allopurinol and benzbromarone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) | Baseline up to 48-weeks
  Recommended phase II dose (RP2D)

SECONDARY OUTCOMES:
The incidence of adverse events (AEs) | Baseline up to 96-weeks
  Number of participants with adverse events (AE) and/or severe adverse events (SAE) and/or abnormal laboratory examination indicators.
The severity of adverse events (AEs) | Baseline up to 96-weeks
  The severity of adverse events (AEs) as assessed by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.
The severity of severe adverse events (SAEs) | Baseline up to 96-weeks
  The severity of severe adverse events (SAEs) as assessed by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.
The severity of abnormal laboratory examination indicators | Baseline up to 96-weeks
  The severity of abnormal laboratory examination indicators as assessed by Common Terminology Criteria for Adverse Events (CTCAE) 5.0.

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing University Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - The Affiliated Hospital of Xuzhou Medical University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital Of Soochow University, Suzhou, Jiangsu
  - Jinzhou Central Hospital, Wuxi, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Shanghai Huashan Hospital, Shanghai, Shanghai Municipality
  - Tongji hospital of Tongji University, Shanghai, Shanghai Municipality
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Institute of Dematology & Blood diseases Hospital, Tianjin, Tianjin Municipality
  - Xinjiang Uygur Autonomous Region People's Hospital, Ürümqi, Xinjiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang